CLINICAL TRIAL: NCT01346150
Title: A Retrospective and Cross-Sectional Analysis of Patients Treated for SCID Since January 1,1968 (RDCRN PIDTC-6902)
Brief Title: Patients Treated for SCID (1968-Present)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Primary Immune Deficiency Treatment Consortium (PIDTC) (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT RDCRN PIDTC-6902
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: SCID; ADA-SCID; XSCID; Leaky SCID; Omenn Syndrome; Reticular Dysgenesis
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency; X-Linked Combined Immunodeficiency Diseases; Severe Combined Immunodeficiency; Reticular dysgenesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biospecimens may include blood, other tissues (e.g., buccal swab or brushing), and/or bone marrow.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Stratum A -Typical SCID: Typical Severe Combined Immunodeficiency (SCID), Adenosine Deaminase-Deficient ADA SCID, and X-linked SCID (XSCID) who received a transplant
- Stratum B - Atypical SCID: Leaky SCID, Omenn Syndrome, and Reticular Dysgenesis who received a transplant
- Stratum C - SCID w/Non-HCT Treatments: SCID who received Polyethylene Glycol -Adenosine Deaminase Enzyme Replacement Therapy (PEG-ADA ERT) or gene therapy

SUMMARY:
Individuals with a past diagnosis of severe combined immune deficiency (including many cases of "leaky SCID", Omenn syndrome, and reticular dysgenesis) who have undergone blood and marrow transplant, gene therapy, or enzyme replacement in the past may be eligible for this study. The purpose of study is to look backwards at what has already been done in the. Over 800 patients with SCID are expected to be enrolled, making this one of the largest studies ever to describe outcomes for patients with SCID treated at many different hospitals around North America.

DETAILED DESCRIPTION:
One of the most important components of this study is the "cross sectional" aspect. Patients who have received their treatments (BMT, gene therapy, enzyme replacement) many years ago are asked to come back to the hospital where they were treated. During this visit, additional research bloodwork is drawn, and information is gathered regarding long-term transplant outcomes such as infections, graft-versus-host disease, autoimmune diseases, and quality of life. This will allow PIDTC researchers to better understand long-term outcomes from procedures that occurred many years ago (sometimes over 30 years ago). This will help researchers to best design new treatments and clinical trials in the future for children with SCID.

ELIGIBILITY:
Inclusion Criteria:

Strata A, B, and C (Part 1 - Retrospective Study)-

* Individuals with Severe Combined Immune Deficiency (SCID) diagnosis who:

  --were treated at a location participating in this consortium from 1968 until present, and

  --are not enrolled in RDCRN PIDTC-6901 (ClinicalTrials.gov ID: NCT01186913).
* Subjects who received HCT/GT/ERT prior to the present date are eligible for the retrospective study. The enrollment criteria for subjects who died prior to definitive therapy are the same as for Strata A, B and C.

Stratum A, Typical SCID:

* Individuals who meet the following inclusion criteria and who received HCT are eligible for enrollment into Stratum A of the study:

  * Absence or very low number of T cells (CD3 T cells < 300/microliter), and no or very low T cell function (< 10% of lower limit of normal) as measured by response to phytohemagglutinin (PHA) or cells of maternal origin present.
  * If maternal cells are present but the patient does not meet criteria for very low T cell function as defined, the assigned reviewers for the potential subject, and if necessary, the full PID-SCID RP will review the laboratory report to determine if criteria of maternal engraftment are met for Protocol 6902.
  * Laboratory report of testing for maternal engraftment is required, for evaluation by the PID-SCID RP.

Stratum B, Leaky SCID, Omenn Syndrome, Reticular Dysgenesis:

Individuals who meet the following criteria are eligible for enrollment into Stratum B of the study:

Leaky SCID-

* Maternal lymphocytes tested for and not detected and,
* Either one or both of the following (a,b):

  a) < 50% of lower limit of normal T cell function (as measured by response to PHA OR < 50% of lower limit of normal T cell function as measured by response to CD3/CD28 antibody, b) Absent or < 30% lower limit of normal proliferative responses to candida and tetanus toxoid antigens postvaccination or exposure,
* AND at least one of the following (a through e):

  1. Reduced number of CD3 T cells,
  2. > 80% of CD3+ or CD4 T cells are CD45RO+,
* AND/OR >80% of CD3+ or CD4+ T cells are,CD62L negative,
* AND/OR >50% of CD3+ or CD4+ T cells express HLA-DR (at < 4 years of age),
* AND/OR are oligoclonal T cells. c) Hypomorphic mutation in IL2RG in a male, or homozygous hypomorphic mutation or compound heterozygosity with at least one hypomorphic mutation in an autosomal SCID-causing gene.

  d) Low TRECs and/or the percentage of CD4+/45RA+/CD31+ or CD4+/45RA+/CD62L+ cells is below the lower limit of normal.

  e) Functional testing in vitro supporting impaired, but not absent, activity of the mutant protein,
  * AND does not meet criteria for Omenn Syndrome,
  * AND does not have known selective loss of lymphocytes, Ataxia- Telangiectasia, or congenital heart defect associated with lymphopenia, unless a SCID genotype is also present.

Omenn Syndrome (OS):

* Generalized skin rash,
* Maternal engraftment tested for and not detected,
* Absent or low (up to 30% of normal) T cell proliferation to antigens to which the patient has been exposed.
* If the proliferation to antigen was not performed, but at least 4 of the following 10 supportive criteria, at least one of which must be among those marked with an asterisk (*) are present, the patient is eligible: hepatomegaly; splenomegaly; lymphadenopathy; elevated IgE; elevated absolute eosinophil count; *oligoclonal T cells measured by CDR3 length or flow cytometry >80% of CD4+ T cells are CD45RO+ ;*proliferation to PHA is reduced <50% of lower limit of normal or SI <30; *proliferative response in mixed leukocyte reaction is reduced to increment cpm < 20% or SI <20; hypomorphic mutation to SCID causing gene; low TRECs and/or percentage of CD 4+/ RA+/CD31+; or CD4+/RA+/CD62L+ cells below the lower limit of normal.

Reticular Dysgenesis (RD):

* Absence or very low number of T cells (CD3 T cells <300/microliter),
* No or very low (<10% of lower limit of normal) T cell function (as measured by response to phytohemagglutinin (PHA),
* Severe congenital neutropenia (absolute neutrophil count <200/microliter),
* AND at least one of the following:

  * Sensorineural deafness and/or absence of granulopoiesis at bone marrow examination and/or a deleterious AK2 mutation,
  * absence of granulopoiesis on bone marrow examination; a pathogenic mutation in the adenylate kinase 2 (AK2) gene identified.

Stratum C, SCID with Non-HCT Treatments:

-Individuals who meet the following criteria and were treated with PEG-ADA or gene therapy with autologous modified cells are eligible for enrollment into Stratum C (SCID with non-HCT treatments) of the study-

- Any SCID patient previously treated with a thymus transplant (includes intention to treat with HCT, as well as PEG-ADA ERT or gene therapy).

Strata A, B, and C (Part 2 - Cross-Sectional Study):

Patient inclusion criteria for the cross sectional study: Eligibility for Strata A, B and C are the same as for the retrospective study except that all the patients in the cross-sectional study are currently surviving and are at least 2 years post the most recent class of therapy.

Exclusion Criteria:

Parts 1 and 2 - Retrospective and Cross-Sectional Studies -

* Lack of appropriate testing to rule out HIV infection after 1997 (p24 antigen or more sensitive) or other cause of secondary immunodeficiency,
* Presence of DiGeorge syndrome,
* Most patients with other PIDs such as nucleoside phosphorylase deficiency, ZAP70 deficiency, CD40 ligand deficiency, NEMO deficiency, XLP, cartilage hair hypoplasia or ataxia telangiectasia will not meet the inclusion criteria for Stratum A, B, or C above; however, a patient with one of the above may meet the inclusion criteria for Stratum B and if so will be included-

  * MHC Class I and MHC Class II antigen deficiency are excluded,
  * Metabolic conditions that imitate SCID or related disorders such as folate transporter deficiency, severe zinc deficiency, transcobalamin deficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with diagnosis of SCID or SCID variants treated at Participating Consortium Centers from 1968-Present
Sampling Method: Non-Probability Sample
Enrollment: 1007 (Estimated)
Dates: Start 2011-05-15 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Retrospective Study - Part 1 | 1, 5, 10, 20, >20 years
  Overall survival
Cross-Sectional Study - Part 2 | 2 to > 20 years
  Full immune reconstitution

SECONDARY OUTCOMES:
Retrospective Study Part 1 | 1 year to > 20 years
  Immune reconstitution and clinical outcomes
Retrospective Study - Part 1 | 3 months to >20 years
  Engraftment
Cross-Sectional Study - Part 2 | 2 to >20 years
  Current state of lineage-specific chimerism
Cross-Sectional Study - Part 2 | 2 to >20 years
  Current status of health

CONTACTS AND LOCATIONS:
Overall Officials: Elie Haddad, MD, PhD, Study Chair — University of Montréal, CHU Sainte-Justine; Richard J. O'Reilly, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Morton J. Cowan, MD, Study Chair — University of California, San Francisco
Locations (36):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA: Division of Pediatric Hematology/Oncology, Los Angeles, California
  - Lucile Salter Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California San Francisco Children's Hospital, San Francisco, California
  - Children's Hospital Denver:Center for Cancer and Blood Disorders, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta/Emory University School of Medicine, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital/Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - NIH Clinical Center Genetic Immunotherapy Section, Bethesda, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - SSM Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University St Louis Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center: Department of Pediatrics, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center: Department of Pediatrics, New York, New York
  - Duke University Medical Center: Department of Pediatrics, Division of Allergy/Immunology, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University: Pediatric Hematology/Oncology, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center/University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center: Clinical Research Division and Pediatric Stem Cell Transplantation Center, Seattle, Washington
  - University of Wisconsin/ American Family Children's Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - CHU St. Justine, Montreal, Quebec

REFERENCES:
- [Background] Griffith LM, Cowan MJ, Kohn DB, Notarangelo LD, Puck JM, Schultz KR, Buckley RH, Eapen M, Kamani NR, O'Reilly RJ, Parkman R, Roifman CM, Sullivan KE, Filipovich AH, Fleisher TA, Shearer WT. Allogeneic hematopoietic cell transplantation for primary immune deficiency diseases: current status and critical needs. J Allergy Clin Immunol. 2008 Dec;122(6):1087-96. doi: 10.1016/j.jaci.2008.09.045. Epub 2008 Nov 6. PMID 18992926
- [Result] Pai SY, Logan BR, Griffith LM, Buckley RH, Parrott RE, Dvorak CC, Kapoor N, Hanson IC, Filipovich AH, Jyonouchi S, Sullivan KE, Small TN, Burroughs L, Skoda-Smith S, Haight AE, Grizzle A, Pulsipher MA, Chan KW, Fuleihan RL, Haddad E, Loechelt B, Aquino VM, Gillio A, Davis J, Knutsen A, Smith AR, Moore TB, Schroeder ML, Goldman FD, Connelly JA, Porteus MH, Xiang Q, Shearer WT, Fleisher TA, Kohn DB, Puck JM, Notarangelo LD, Cowan MJ, O'Reilly RJ. Transplantation outcomes for severe combined immunodeficiency, 2000-2009. N Engl J Med. 2014 Jul 31;371(5):434-46. doi: 10.1056/NEJMoa1401177. PMID 25075835
- [Result] Shearer WT, Dunn E, Notarangelo LD, Dvorak CC, Puck JM, Logan BR, Griffith LM, Kohn DB, O'Reilly RJ, Fleisher TA, Pai SY, Martinez CA, Buckley RH, Cowan MJ. Establishing diagnostic criteria for severe combined immunodeficiency disease (SCID), leaky SCID, and Omenn syndrome: the Primary Immune Deficiency Treatment Consortium experience. J Allergy Clin Immunol. 2014 Apr;133(4):1092-8. doi: 10.1016/j.jaci.2013.09.044. Epub 2013 Nov 28. PMID 24290292
- [Result] Haddad E, Allakhverdi Z, Griffith LM, Cowan MJ, Notarangelo LD. Survey on retransplantation criteria for patients with severe combined immunodeficiency. J Allergy Clin Immunol. 2014 Feb;133(2):597-9. doi: 10.1016/j.jaci.2013.10.022. Epub 2013 Dec 10. No abstract available. PMID 24331379
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Kohn DB, Puck JM, Shearer WT, Burroughs LM, Torgerson TR, Decaluwe H, Haddad E; workshop participants. Primary Immune Deficiency Treatment Consortium (PIDTC) update. J Allergy Clin Immunol. 2016 Aug;138(2):375-85. doi: 10.1016/j.jaci.2016.01.051. Epub 2016 Apr 22. PMID 27262745
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Kohn DB, Puck JM, Pai SY, Ballard B, Bauer SC, Bleesing JJ, Boyle M, Brower A, Buckley RH, van der Burg M, Burroughs LM, Candotti F, Cant AJ, Chatila T, Cunningham-Rundles C, Dinauer MC, Dvorak CC, Filipovich AH, Fleisher TA, Bobby Gaspar H, Gungor T, Haddad E, Hovermale E, Huang F, Hurley A, Hurley M, Iyengar S, Kang EM, Logan BR, Long-Boyle JR, Malech HL, McGhee SA, Modell F, Modell V, Ochs HD, O'Reilly RJ, Parkman R, Rawlings DJ, Routes JM, Shearer WT, Small TN, Smith H, Sullivan KE, Szabolcs P, Thrasher A, Torgerson TR, Veys P, Weinberg K, Zuniga-Pflucker JC; workshop participants. Primary Immune Deficiency Treatment Consortium (PIDTC) report. J Allergy Clin Immunol. 2014 Feb;133(2):335-47. doi: 10.1016/j.jaci.2013.07.052. Epub 2013 Oct 15. PMID 24139498
- [Result] Dvorak CC, Cowan MJ, Logan BR, Notarangelo LD, Griffith LM, Puck JM, Kohn DB, Shearer WT, O'Reilly RJ, Fleisher TA, Pai SY, Hanson IC, Pulsipher MA, Fuleihan R, Filipovich A, Goldman F, Kapoor N, Small T, Smith A, Chan KW, Cuvelier G, Heimall J, Knutsen A, Loechelt B, Moore T, Buckley RH. The natural history of children with severe combined immunodeficiency: baseline features of the first fifty patients of the primary immune deficiency treatment consortium prospective study 6901. J Clin Immunol. 2013 Oct;33(7):1156-64. doi: 10.1007/s10875-013-9917-y. Epub 2013 Jul 2. PMID 23818196
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Puck JM, Buckley RH, Candotti F, Conley ME, Fleisher TA, Gaspar HB, Kohn DB, Ochs HD, O'Reilly RJ, Rizzo JD, Roifman CM, Small TN, Shearer WT; Workshop Participants. Improving cellular therapy for primary immune deficiency diseases: recognition, diagnosis, and management. J Allergy Clin Immunol. 2009 Dec;124(6):1152-60.e12. doi: 10.1016/j.jaci.2009.10.022. PMID 20004776
- [Result] Kohn DB, Hershfield MS, Puck JM, Aiuti A, Blincoe A, Gaspar HB, Notarangelo LD, Grunebaum E. Consensus approach for the management of severe combined immune deficiency caused by adenosine deaminase deficiency. J Allergy Clin Immunol. 2019 Mar;143(3):852-863. doi: 10.1016/j.jaci.2018.08.024. Epub 2018 Sep 5. PMID 30194989
- [Result] Miggelbrink AM, Logan BR, Buckley RH, Parrott RE, Dvorak CC, Kapoor N, Abdel-Azim H, Prockop SE, Shyr D, Decaluwe H, Hanson IC, Gillio A, Davila Saldana BJ, Eibel H, Hopkins G, Walter JE, Whangbo JS, Kohn DB, Puck JM, Cowan MJ, Griffith LM, Haddad E, O'Reilly RJ, Notarangelo LD, Pai SY. B-cell differentiation and IL-21 response in IL2RG/JAK3 SCID patients after hematopoietic stem cell transplantation. Blood. 2018 Jun 28;131(26):2967-2977. doi: 10.1182/blood-2017-10-809822. Epub 2018 May 4. PMID 29728406
- [Result] Haddad E, Logan BR, Griffith LM, Buckley RH, Parrott RE, Prockop SE, Small TN, Chaisson J, Dvorak CC, Murnane M, Kapoor N, Abdel-Azim H, Hanson IC, Martinez C, Bleesing JJH, Chandra S, Smith AR, Cavanaugh ME, Jyonouchi S, Sullivan KE, Burroughs L, Skoda-Smith S, Haight AE, Tumlin AG, Quigg TC, Taylor C, Davila Saldana BJ, Keller MD, Seroogy CM, Desantes KB, Petrovic A, Leiding JW, Shyr DC, Decaluwe H, Teira P, Gillio AP, Knutsen AP, Moore TB, Kletzel M, Craddock JA, Aquino V, Davis JH, Yu LC, Cuvelier GDE, Bednarski JJ, Goldman FD, Kang EM, Shereck E, Porteus MH, Connelly JA, Fleisher TA, Malech HL, Shearer WT, Szabolcs P, Thakar MS, Vander Lugt MT, Heimall J, Yin Z, Pulsipher MA, Pai SY, Kohn DB, Puck JM, Cowan MJ, O'Reilly RJ, Notarangelo LD. SCID genotype and 6-month posttransplant CD4 count predict survival and immune recovery. Blood. 2018 Oct 25;132(17):1737-1749. doi: 10.1182/blood-2018-03-840702. Epub 2018 Aug 28. PMID 30154114
- [Result] Dvorak CC, Haddad E, Buckley RH, Cowan MJ, Logan B, Griffith LM, Kohn DB, Pai SY, Notarangelo L, Shearer W, Prockop S, Kapoor N, Heimall J, Chaudhury S, Shyr D, Chandra S, Cuvelier G, Moore T, Shenoy S, Goldman F, Smith AR, Sunkersett G, Vander Lugt M, Caywood E, Quigg T, Torgerson T, Chandrakasan S, Craddock J, Davila Saldana BJ, Gillio A, Shereck E, Aquino V, DeSantes K, Knutsen A, Thakar M, Yu L, Puck JM. The genetic landscape of severe combined immunodeficiency in the United States and Canada in the current era (2010-2018). J Allergy Clin Immunol. 2019 Jan;143(1):405-407. doi: 10.1016/j.jaci.2018.08.027. Epub 2018 Sep 5. PMID 30193840
- [Derived] Rayes A, Logan BR, Liu X, Dara J, Buckley RH, Oved JH, Kapoor N, Kapadia M, Chandra S, Martinez CA, Bunin N, Chandrakasan S, Chen K, Bednarski JJ, Haines HL, Eissa H, Talano JM, Keller MD, Ebens CL, Chaudhury S, Shereck EB, Aquino VM, Knutsen AP, Alexander JL, Gillio AP, Chellapandian D, Shah AJ, Miller HK, Vander Lugt MT, Seroogy CM, Dorsey MJ, Mousallem T, Parrott RE, O'Reilly RJ, Aguayo-Hiraldo PI, Prockop SE, Davila Saldana BJ, Thakar MS, Burroughs LM, Torgerson TR, Leiding JW, Marsh RA, Griffith LM, Pulsipher MA, Kohn DB, Notarangelo LD, Cowan MJ, Puck JM, Cuvelier GDE, Heimall J, Haddad E, Pai SY, Dvorak CC. Outcomes Following Matched Sibling Donor Transplantation for Severe Combined Immunodeficiency: A Report from the PIDTC. Blood Adv. 2025 Nov 25:bloodadvances.2025016812. doi: 10.1182/bloodadvances.2025016812. Online ahead of print. PMID 41289158
- [Derived] Cuvelier GDE, Logan BR, Prockop SE, Buckley RH, Kuo CY, Griffith LM, Liu X, Yip A, Hershfield MS, Ayoub PG, Moore TB, Dorsey MJ, O'Reilly RJ, Kapoor N, Pai SY, Kapadia M, Ebens CL, Forbes Satter LR, Burroughs LM, Petrovic A, Chellapandian D, Heimall J, Shyr DC, Rayes A, Bednarski JJ, Chandra S, Chandrakasan S, Gillio AP, Madden L, Quigg TC, Caywood EH, Davila Saldana BJ, DeSantes K, Eissa H, Goldman FD, Rozmus J, Shah AJ, Vander Lugt MT, Thakar MS, Parrott RE, Martinez C, Leiding JW, Torgerson TR, Pulsipher MA, Notarangelo LD, Cowan MJ, Dvorak CC, Haddad E, Puck JM, Kohn DB. Outcomes following treatment for ADA-deficient severe combined immunodeficiency: a report from the PIDTC. Blood. 2022 Aug 18;140(7):685-705. doi: 10.1182/blood.2022016196. PMID 35671392
- See also: Primary Immune Deficiency Treatment Consortium (PIDTC) — https://www.rarediseasesnetwork.org/cms/pidtc
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: National Center for Advancing Translational Sciences (NCATS) — https://ncats.nih.gov/